CLINICAL TRIAL: NCT00464204
Title: Effects of Voluven on Hemodynamics and Tolerability of Enteral Nutrition in Patients With Severe Sepsis
Acronym: CRYSTMAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-HE06-01; 2006-004350-25 (EudraCT Number)
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — HES 130-0.4; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voluven® Arm (Experimental)
  Interventions: Drug: 6 % Hydroxyethylstarch 130/0.4 = "Voluven®"
- 0.9 % NaCl (Active Comparator)
  Interventions: Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: 6 % Hydroxyethylstarch 130/0.4 = "Voluven®" — Voluven® was administered intravenously. Voluven® rates were not to exceed 50 mL/kg/day on the first day and 25 mL/kg/day on the second to fourth days, according to patient needs.
  Other Names: Voluven®
  Arms: Voluven® Arm
Drug: 0.9 % NaCl — NaCl 0.9 % was administered intravenously. NaCl 0.9% rates were not to exceed 50 mL/kg/day on the first day and 25 mL/kg/day from the second to the fourth day, according to patient needs.
  Arms: 0.9 % NaCl

SUMMARY:
The rapidity and the quality of fluid resuscitation in patients with severe sepsis are important factors for the prevention of secondary multi-organ failure. Vascular filling may also have an impact on tolerability of enteral nutrition. The earliness and quantity of calories provided by enteral nutrition may have an impact on morbidity and mortality. This study will asses the effects of volume expansion on hemodynamics and tolerability of enteral nutrition in patients with severe sepsis. A Data Monitoring Committee will review regularly safety data of the study.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Requirement for fluid resuscitation

Exclusion Criteria:

* serum creatinine > 300µmol/L
* Chronic renal failure
* Anuria lasting more than 4 hours
* Requirement for renal support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Guidet, Prof., MD, Study Chair — Hôpital St Antoine, Réanimation Médicale
Locations (24):
- France (21):
  - Hôpital Sud, Unité de Réanimation Médicale, Amiens
  - Centre Hospitalier d'Avignon, Service de Réanimation Polyvalente, Avignon
  - Centre Hospitalier de Belfort-Montbéliard, Service de Réanimation et Maladies Infectieuses, Site de Belfort, Belfort
  - CHU de Bicêtre, Dpt d'Anesthésie Réanimation Chir., Bicêtre
  - Hôpital Avicenne, Service de Réanimation, Bobigny
  - Centre Hospitalier Fleyriat, Service de Réanimation Polyvalente, Bourg-en-Bresse
  - CH Manchester, Service de Réanimation Polyvalente, Charleville-Mézières
  - CH Sud Francilien, Site Gilles de Corbeil, Réanimation Polyvalente, Corbeil-Essonnes
  - CHU de Dijon - Hôpital du Bocage Service de Réanimation Médicale, Dijon
  - CH Meaux, Service de Réanimation, Meaux
  - Centre Hospitalier de Metz, Réa Polyvalente, Metz
  - Hôpital Lapeyronie / CHU Montpellier, Département d'Anesthésie Réanimation, Montpellier
  - Hôpital Central, Service Anesthésie-Réanimation, Chirurgicale CHU, Nancy
  - CHU Nîmes, Service de Réanimation, Division Anesthésie-Réa Douleur Urgence, Groupe Hospitalo-Universitaire Caremeau,, Nîmes
  - Hôpital de la Source, Réanimation Polyvalente, Orléans
  - Hôpital St Louis, Département Anesthésie et Réanimation Chirurgicale, Paris
  - Hôpital Saint-Joseph, Service de Réanimation Polyvalente, Paris
  - Hôpital St Antoine, Réanimation Médicale, Paris
  - CH Roanne, Service de Réanimation, Roanne
  - CHI Poissy - St Germain en Laye, Site de St Germain en Laye, Saint-Germain-en-Laye
  - Hôpital Civil de Strasbourg, Service de Réanimation Médicale, Strasbourg
- Germany (3):
  - Klinik und Poliklinik für Anästhesiologie und Intensivtherapie - Universitätsklinikum Leipzig AöR, Leipzig
  - Klinik und Poliklinik für Anästhesiologie und operative Intensivmedizin der Westf. Wilhelms-Universität, Münster
  - Universitätsklinikum Tübingen, Klinik für Anästhesiologie und Intensivmedizin, Tübingen

REFERENCES:
- [Derived] Guidet B, Martinet O, Boulain T, Philippart F, Poussel JF, Maizel J, Forceville X, Feissel M, Hasselmann M, Heininger A, Van Aken H. Assessment of hemodynamic efficacy and safety of 6% hydroxyethylstarch 130/0.4 vs. 0.9% NaCl fluid replacement in patients with severe sepsis: the CRYSTMAS study. Crit Care. 2012 May 24;16(3):R94. doi: 10.1186/cc11358. PMID 22624531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 24 intensive care units of hospitals in France and Germany from July 2007 until February 2010 and were followed up until May 2010.
Pre-assignment Details: Participants were screened in intensive care units of the participating study sites in France and Germany.
Groups:
- Voluven® Arm: 6 % Hydroxyethylstarch 130/0.4; Voluven® rates were not to exceed 50 mL/kg/day on the first days and 25 mL/kg/day from the second to the fourth day
- NaCl 0.9 % Arm: NaCl 0.9 %; NaCl 0.9 % rates were not to exceed 50 mL/kg/day on the first day and 25 mL/kg/day from the second to the fourth day
Period: Overall Study
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Started | 100 | 96
Completed Treatment | 81 | 83
Day 30 Follow-up Performed | 89 | 83
Day 90 Follow-up Performed | 69 | 74
Withdrawal Due to Discharge From ICU | 18 | 11
Completed | 51 (Completed=no withdrawal until day 8.) | 64 (Completed=no withdrawal until day 8.)
Not Completed | 49 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm | Total
Number analyzed (Participants) | 100 | 96 | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 65.8 (15.4) | 65.9 (14.7) | 65.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 64 | 57 | 121
Region of Enrollment [Number; unit: participants]
  France | 87 | 84 | 171
  Germany | 13 | 12 | 25
Origin of sepsis [Number; unit: participants] — Multiple origins of sepsis could be reported for a single patient.
  participants
    Lungs | 53 | 58 | 111
    Abdomen | 24 | 18 | 42
    Urogenital | 8 | 14 | 22
    Skin, bone and soft tissue | 6 | 4 | 10
    Other | 5 | 2 | 7
    Unknown | 4 | 2 | 6
    Neurological system | 3 | 2 | 5
    Ears-nose-throat system | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Amount of Study Drug Required to Achieve Initial Hemodynamic Stabilization
Description: Initial hemodynamic stabilization (HDS) was defined as normalization of mean arterial pressure (MAP) and at least two of the three parameters central venous pressure (CVP), urine output and central venous oxygen saturation and maintaining this normalization over a period of four hours, with no increase in the infusion of vasopressors, or ionotropic therapy and with no more than 1 L of additional study drug administration within these four hours.
Time Frame: until hemodynamic stabilization (up to 48 hours)
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 88 | 86
Milliliter | 1379 (886) | 1709 (1164)
Statistical Analysis 1: Comparison: Voluven® Arm vs NaCl 0.9 % Arm; Null-hypothesis: The amount of study drug required to achieve initial hemodynamic stabilization in patients treated with Voluven® is higher than or equal to this amount in patients treated with NaCl. Alternative hypothesis: The amount of study drug required to achieve initial hemodynamic stabilization is lower in patients treated with Voluven® than in patients treated with NaCl; Test type: Superiority or Other; p = 0.0185, t-test, 1 sided — One-sided t-test assuming unequal variances (as variances were significantly different between treatment groups).No multiple comparisons were made. A priori threshold for statistical significance for the confirmatory analysis on FAS: 0.025 one-sided; Mean Difference (Final Values) = -331, 95% CI 2-sided [-640 to -21], Standard Deviation 1033 — Considered difference: Voluven® minus NaCl 0.9 %

2. Secondary Outcome: Time From Start of Fluid Resuscitation With Study Drug to the Initial Hemodynamic Stabilization
Description: Time from start of fluid resuscitation with study drug to the initial hemodynamic stabilization
Time Frame: until hemodynamic stabilization (up to 48 hours)
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 88 | 86
Hours | 11.8 (10.1) | 14.3 (11.1)

3. Secondary Outcome: Quantity of Study Drug in 4 Days
Description: Total quantity of study drug infused over four consecutive days in the ICU
Time Frame: 4 days
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 88 | 86
Milliliter | 2615 (1499) | 2788 (1799)

4. Secondary Outcome: Time From Start of Study Drug to Start of Enteral Nutrition in the Subgroup of Patients Who Received Enteral Nutrition
Description: Time from start of fluid resuscitation with study drug to start of enteral nutrition.
Time Frame: Until start of enteral nutrition (up to 48 hours)
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 62 | 67
Hours | 24.6 (32.7) | 26.9 (33.8)

5. Secondary Outcome: Time From Start of Fluid Resuscitation With Study Drug to Start of Enteral Nutrition After Hemodynamic Stabilization
Description: Administration of enteral nutrition before initial hemodynamic stabilization was ignored in this analysis.
Time Frame: up to 48 hours
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 62 | 67
Hours | 25.9 (32.1) | 27.6 (33.6)

6. Secondary Outcome: Total Amount of Enteral Calories During the First Seven Days of Enteral Nutrition
Description: This amount will be calculated from start of enteral nutrition until 7 am of day 8
Time Frame: 7 days
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 62 | 67
kcal | 6877 (5008) | 7429 (4381)

7. Secondary Outcome: Length of Stay in the Intensive Care Unit (ICU)
Description: Length of stay was analysed in two approaches. First, it was calculated and analysed only for patients who did not die before end of study of the individual patient. As a sensitivity analysis, the analysis was carried out including patients who died with the maximum possible length of stay (i.e., the worst possible value).
Time Frame: Until discharge from ICU (up to day 90)
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization.
  Calculated for patients who did not die before end of study of the individual patient
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 58 | 61
Days | 15.4 (11.1) | 20.2 (22.2)

8. Secondary Outcome: Length of Stay in the ICU
Description: Length of stay was analysed in two approaches. First, it was calculated and analysed only for patients who did not die before end of study of the individual patient. As a sensitivity analysis, the analysis was carried out including patients who died with the maximum possible length of stay (i.e., worst possible value).
Time Frame: Until discharge from ICU (up to Day 90)
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization.
  Imputed with the longest possible duration for patients who died before end of the study of the individual patient.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 88 | 86
Days | 40.0 (36.5) | 39.6 (36.3)

9. Secondary Outcome: Length of Stay in the Hospital
Description: as for outcome 7
Time Frame: Until discharge from hospital (up to day 90)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 58 | 61
Days | 37.7 (26.5) | 42.7 (31.6)

10. Secondary Outcome: Length of Stay in the Hospital
Description: as for outcome 7
Time Frame: Until discharge from hospital (up to Day 90)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 88 | 86
Days | 56.1 (33.5) | 56.9 (34.7)

11. Secondary Outcome: Area Under the Curve (AUC) of Sepsis-related Organ Failure Assessment (SOFA) Score Per Day From Screening to Day 4
Description: The Sepsis-related Organ Failure Assessment (SOFA) score in this study is reported for entire days, not for exact time points on a day. Potentially, more than one SOFA score may be available for the same day. In this case, the mean of the respective total scores was used for that day for calculation of Area Under the Curve (AUC).
  The SOFA score includes sub-scores for Respiration, Coagulation, Liver, Cardiovascular, Central Nervous System and Renal function and may range from 0 (worst outcome) to 4 (best outcome).
Time Frame: From Screening to Day 4
Population: Full analysis set (FAS) = all randomized patients treated with study drug who reached hemodynamic stabilization
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 82 | 74
Scores on a scale | 6.9 (3.3) | 7.6 (3.1)

12. Other Pre Specified Outcome: Mortality
Description: Mortality was reported for the time period from Screening until the end of follow-up.
Time Frame: From Screening to end of Follow-up
Population: Treated population (TRT) = all randomized patients treated with study drug. Two patients in the Voluven® arm died due to non-treatment emergent SAEs.
Measure: Number; unit: Participants
Groups:
- Voluven® Arm: 6 % Hydroxyethylstarch 130/0.4 Voluven® rates were not to exceed 50 mL/kg/day on the first day and 25 mL/kg/day from the second to the fourth day.
- NaCl 0.9 % Arm: NaCl 0.9 % NaCl 0.9 % rates were not to exceed 50 mL/kg/day on the first day and 25 mL/kg/day from the second to the fourth day
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 100 | 96
Participants
  From screening until (and including) Day 28 | 31 | 24
  From screening until end of follow-up | 40 | 32

13. Other Pre Specified Outcome: Changes in Renal Function: 1. Acute Renal Failure (ARF) at Any Time After Screening
Description: Acute Renal Failure (ARF) was defined as a two fold increase in serum concentration over the value at screening at any time after screening.
Time Frame: From screening to end of follow-up (up to day 90)
Population: Treated population (TRT) = all randomized patients treated with study drug. Patients without ARF were excluded from analysis if they had no creatinine value at Screening or no post-screening creatinine value.
Measure: Number; unit: Participants
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 98 | 95
Participants | 24 | 19

14. Other Pre Specified Outcome: Changes in Renal Function: 2. Acute Kidney Injury Network (AKIN) Classification
Description: Acute Kidney Injury Network (AKIN) Classification in this study is based on serum creatinine values and renal replacement therapy, i.e. ignoring criteria based on urine output, as fulfilment of urine output criteria cannot be determined from the data collected in the study. AKIN ranges from stage 1 to stage 3 (worst outcome). Stages differ in serum creatinine increase. Stage 1: Increase ≥ 0.3mg/dL or ≥ 150%-200% from reference; Stage 2: Increase ≥ 200%-300% from reference; Stage 3: Increase >300% from reference with an acute increase of at least 0.5mg/dL or renal replacement therapy.
Time Frame: From screening to end of follow-up
Population: Treated population (TRT) = all randomized patients treated with study drug
Measure: Number; unit: Participants
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 100 | 96
Participants
  None | 52 | 52
  AKIN Stage 1 | 21 | 21
  AKIN Stage 2 | 5 | 6
  AKIN Stage 3 | 22 | 17

15. Other Pre Specified Outcome: Changes in Renal Function: 3. Risk, Injury, Failure, Loss, End-stage Kidney Disease (RIFLE) Classification
Description: Risk, Injury, Failure, Loss, End-stage kidney disease (RIFLE) Classification in this study is based on serum creatinine values and renal replacement therapy, i.e. ignoring criteria based on urine output, as fulfilment of urine output criteria cannot be determined from the data collected in the study.
  RIFLE comprises five categories: Risk (R), Injury (I), Failure (F), Loss (L), End-stage kidney disease (E) (worst outcome). R, I and F are based on increase in serum creatinine. L and E are based on administration of renal replacement therapy.
Time Frame: From screening to end of follow-up
Population: Treated population (TRT) = all randomized patients treated with study drug
Measure: Number; unit: Participants
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Number analyzed (Participants) | 100 | 96
Participants
  None | 77 | 73
  Risk | 13 | 11
  Injury | 4 | 5
  Failure | 5 | 7
  Loss | 1 | 0
  End-stage kidney disease | 0 | 0

ADVERSE EVENTS:
Description: Regular assessment by Pharmacovigilance and Safety Assessor
Arm/Group | Voluven® Arm | NaCl 0.9 % Arm
Serious Adverse Events (participants affected / at risk) | 53/100 | 44/96
Other Adverse Events (participants affected / at risk) | 99/100 | 95/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voluven® Arm (N=100) | NaCl 0.9 % Arm (N=96)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute right ventricular failure (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 6
Cardiac tamponade (Cardiac disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 1
Condition aggravated (General disorders) | 4 | 0
Multi-organ failure (General disorders) | 7 | 5
Oedema due to cardiac disease (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 9 | 8
Haemodilution (Injury, poisoning and procedural complications) | 8 | 9
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Blood chloride increased (Investigations) | 0 | 1
Venous oxygen saturation decreased (Investigations) | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Marasmus (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral disorder (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 0 | 2
Acute pulmonary oedema (Reproductive system and breast disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Withdrawal of life support (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voluven® Arm (N=100) | NaCl 0.9 % Arm (N=96)
Anaemia (Blood and lymphatic system disorders) | 22 | 21
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 4
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 6 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cyanosis (Cardiac disorders) | 0 | 1
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 9 | 9
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Pupils unequal (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 5
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 9 | 16
Diarrhoea (Gastrointestinal disorders) | 17 | 22
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Malaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 15 | 17
Chest pain (General disorders) | 1 | 1
Device breakage (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 3 | 4
Oedema due to cardiac disease (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 4 | 4
Pyrexia (General disorders) | 13 | 3
Cholangiolitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemodilution (Injury, poisoning and procedural complications) | 9 | 10
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Aspiration bronchial (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood bicarbonate increased (Investigations) | 1 | 0
Blood creatine increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 3 | 2
Central venous pressure decreased (Investigations) | 2 | 1
Coagulation test abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Mean arterial pressure decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 2
PO2 decreased (Investigations) | 2 | 0
PO2 increased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 19 | 15
Venous oxygen saturation decreased (Investigations) | 6 | 12
Weight increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 7 | 13
Alkalosis (Metabolism and nutrition disorders) | 16 | 14
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 23 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 3
Hyperlactacidaemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 4
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 29
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 29 | 22
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 3
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 2 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 3
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Myoclonus (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 3 | 12
Anxiety (Psychiatric disorders) | 1 | 3
Confusional state (Psychiatric disorders) | 3 | 1
Delirium (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 4 | 0
Oliguria (Renal and urinary disorders) | 4 | 5
Renal failure (Renal and urinary disorders) | 8 | 6
Renal failure acute (Renal and urinary disorders) | 7 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 33 | 35
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 9 | 8
Hypotension (Vascular disorders) | 35 | 38
Labile hypertension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All investigators agreed that there will be one or more publications describing the study and the results. No center or combination of centers will submit their results for publication separately. Highest recruiting centers and Fresenius Kabi will contribute authors. The writing of the manuscript will be a collaborative effort.